CLINICAL TRIAL: NCT05246527
Title: Acute Effects of Physical Exercise in Patients with Borderline Personality Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Aylin Mehren, Dr., Principal Investigator, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ExBPD
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise condition: cycle on an ergometer with moderate or high intensity Control condition: watching a movie
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): 30 min of cycling on a stationary ergometer, guided by a video of a professional cycling instructor.
  * Half of the patients (n=30) and their respective matched healthy controls (n=30) will perform moderate-intensity exercise: continuous cycling at 64-76% of the individual HRmax).
  * The other half will perform a high-intensity interval training (HIIT) protocol: 5 min warm-up phase, followed by bursts of high-intensity cycling interspersed with varied recovery times (21 min in total), 4 min cool-down. Excluding warm-up and cool-down, intensities will remain >77% of individual HRmax during the whole routine.
  Heart rate will be continuously recorded using a chest strap heart rate monitor and monitored by the patients themselves and the experimenter.
  Interventions: Behavioral: Physical Exercise
- Control condition (Active Comparator): 30 min of watching a documentary about the benefits of physical activity on health. Heart rate will be recorded also during the control condition.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Physical Exercise — 30 min of cycling on an ergometer, moderate or high intensity
  Arms: Exercise
Behavioral: Control Intervention — 30 min of watching a movie
  Arms: Control condition

SUMMARY:
The aim of the proposed project is to investigate the effects of a single session of physical exercise on stress regulation, cognitive and emotional functioning, and associated neurophysiological processes (saliva and blood samples) in patients with borderline personality disorder. A further aim is to identify the optimal exercise intensity (moderate vs. high intensity). The investigatiors expect that acute exercise will lead to positive effects on behavioral and biomarker level.

DETAILED DESCRIPTION:
Background: Borderline personality disorder (BPD) is one of the most common personality disorders, with a lifetime prevalence of up to 5.9% and core symptoms of emotional and behavioral dysregulation, instability in interpersonal relationships, identity disturbances, stress-related dissociation, non-suicidal self-injuries, and suicidal behavior. Treatment mainly consists of psychotherapeutic procedures, frequently supplemented by pharmacotherapy to reduce specific symptoms such as affective and cognitive dysregulation. Besides possible adverse effects from medication, both, psychotherapy and medication do not lead to a complete remission of BPD. Previous studies point towards a positive influence of physical exercise on BPD symptoms and related neurobiological processes, while to our knowledge no study has investigated the effects of exercise in patients with BPD yet.

Objectives: To investigate the effects of a single session of physical exercise on stress regulation, cognitive and emotional functioning, and associated neurophysiological processes in patients with borderline personality disorder. A further aim is to identify the optimal exercise intensity (moderate vs. high intensity).

Hypotheses: The investigatiors expect that acute exercise will enhance stress perception and cognitive and emotional functioning, which will be reflected in enhanced behavioral measures and changes on biomarker level. In addition, the investigatiors expect to gather insights regarding the optimal exercise intensity.

Methods: 60 patients with borderline personality disorder and 60 healthy controls will participate in two 30-min experimental conditions on separate days in counterbalanced order (at least 48 hours apart): in the exercise condition, half of the group will cycle on an ergometer with moderate intensity, the other half will perform a high-intensity interval training. Intensities will be calculated based on the individual maximal heart rate measured during a maximal exercise test in a pre-experimental session. In the control condition, all participants will watch a movie. Before and after each condition, they will perform a classic and an emotional version of the Stroop test, in order to assess exercise effects on impulsivity and emotion regulation. To test for exercise effects on stress-related responses, they will further participate in a Stress test 90 min following each condition. The investigatiors will collect saliva and blood samples together with state questionnaires at various study time points to test for effects on peripheral biomarkers related to stress, cognition, and BPD pathology (e.g., cortisol, alpha-amylase, serotonin metabolism, noradrenaline, BDNF).

ELIGIBILITY:
Inclusion Criteria:

* estimated verbal intelligence quotient >80 (MWT-B; Lehrl 2005)
* patients: diagnosis of borderline personality disorder according to DSM-5

Exclusion Criteria:

* neurological disorders
* health conditions interfering with exercise safety, e.g. coronary heart disease
* visual impairments that may interfere with performance of the cognitive tasks
* endocrine disorders, e.g. hyperthyreosis or diabetes mellitus;
* following psychiatric disorders: psychosis or affective disorders with psychotic symptoms, schizophrenia, substance abuse or dependence, autism spectrum disorders, anorexia nervosa;
* healthy controls: BPD, intake of psychotropic drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in cognitive interference | directly before and 10 minutes after exercise and control condition
  classical color-word Stroop task: reaction time difference between congruent and incongruent stimuli, difference between pre- and post-intervention is compared between exercise and control condition
change in subjective stress perception | stress test 90 minutes after exercise and control condition, subjective stress scale are collected before stress test and 0, 10, 20, and 30 minutes after stress test
  Trier social stress test: subjective stress level (visual analogue scale rated from 0=noperceived stress to 9=highest perceived stress), changes between pre-stress and post-stress are compared between exercise and control condition
change in cortisol levels | stress test 90 minutes after exercise and control condition, saliva samples are collected before stress test and 0, 10, 20, and 30 minutes after stress test
  Trier social stress test: cortisol levels measured in saliva; changes between pre-stress and post-stress (cortisol peak expected at 20 minutes after stress test) are compared between exercise and control condition

SECONDARY OUTCOMES:
change in emotional interference | directly before and 15 minutes after exercise and control condition
  emotional Stroop task: reaction time difference between neutral and emotional words, difference between pre- and post-intervention is compared between exercise and control condition
change in affect | directly before and 5 minutes after exercise and control condition, and before stress test and 0, 10, 20, and 30 minutes after stress test
  Positive and Negative Affect Scale (PANAS)
change in alpha-amylase | saliva samples are collected before stress test and 0, 10, 20, and 30 minutes after stress test
  measured in saliva; changes between pre-stress and post-stress are compared between exercise and control condition
change in biomarkers | directly before and 5 minutes after exercise and control condition
  blood samples to measure: serotonin metabolism (e.g., tryptophan metabolism: tryptophan, kynurenine, and kynurenine acid), BDNF, Lactate, Noradrenaline

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided